CLINICAL TRIAL: NCT02861027
Title: Effect of Functional Electrical Stimulation in Gluteus Medius in Rehabilitation After Total Hip Arthroplasty: Randomized Clinical Trial
Brief Title: Effect of Functional Electrical Stimulation in Gluteus Medius in Rehabilitation After Total Hip Arthroplasty
Acronym: EFESGMRTHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Carolina Sant Anna Umpierres, Master Degree, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRioGrande
Record Dates: First submitted 2015-08-19; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: OSTEOARTHRITIS
Keywords: Osteoarthritis; Total hip arthroplasty; Physiotherapy; Functional Electrical Stimulation
MeSH Terms: conditions — Osteoarthritis | interventions — proto-oncogene protein c-fes-fps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PPTHA (Active Comparator): Control Group performs the PPTHA.
  Interventions: Procedure: PPTHA
- FES and PPTHA (Experimental): The Intervention Group performs the PPTHA associated with FES.
  Interventions: Procedure: PPTHA; Procedure: FES and PPTHA

INTERVENTIONS:
Procedure: PPTHA — The control group will receive Protocol Physiotherapeutic Total Hip Arthroplasty (PPTHA), consisting of guidelines on the care and post THA. The PPTHA, is held once a day, for 60 minutes, accompanied by a physiotherapist and has the following composition: 1 day) oral guidance and exercise to strengthen the gluteal muscles and muscles of the thigh, with recommendation for 3 repetitions of 12 movements, for each financial year. Patients are encouraged to sit outside the bed, after the exercises; Day 2) patients perform exercises the first day and begin the March training, with the aid of a Walker or crutches Canadians for the room; Day 3) patients perform exercises and are encouraged to walk in the hallway of the hospital wing. Day 4) reassessment and discharge.
Procedure: FES and PPTHA — The PPTHA associated with FES. The stimulation protocol of FES is performed with the patient positioned in supine position in bed. After cleaning the skin, two electrodes are positioned in the posterolateral region of the thigh in motor point of the medium gluteus muscle. The total time for application of the apparatus 30 min per day totaling more 1 min per day as suggested in specialized references. The intensity is adjusted according to the tolerance of the patient. The apparatus used is wavelength Ibramed Neurodyn Compact.
  Arms: FES and PPTHA

SUMMARY:
Due to the importance of the functions of the gluteus medium, mainly during gait, it becomes essential to strengthening early in the musculature. The association of muscle strengthening with the Functional Electric Stimulation (FES) comes to accelerate stabilization of hip, leading to functional rehabilitation early and improves the quality of life through rehabilitation in social life and activities of daily life. Thus, it becomes a relevant study to assess objectively the implications of FES in muscle strengthening of gluteus medium associated with the Physiotherapy Protocol Total Hip Arthroplasty (PPTHA), through the assessment of motor performance in patients undergoing surgery for Total Hip Arthroplasty (THA), aiming to better rehabilitation strategies for this population.

The objective of the research is to assess the effects of functional rehabilitation through PPTHA associated with FES in the gluteus medium compared only with the PPTHA, in patients undergoing surgery for THA.

The principal hypothesis is that there is difference between the functional rehabilitation of the patients undergoing PPTHA associated with the FES of gluteus medium, after THA and the patients submitted only to PPTHA.

DETAILED DESCRIPTION:
The data collection, evolution and physiotherapy treatment will be carried out on the premises of the Hospital de Clinical de Porto Alegre (HCPA), after approval by the Ethics and Research Committee (ERC) of the institution. The population will consist of patients undergoing surgery for THA at HCPA.

The researchers invite patients that intern consecutively at HCPA, for surgery of THA and fall within the eligibility criteria, to participate in the research. They will be informed about the study, objectives, benefits and potential risks. After the informed consent of the patients and signed the Free and Informed Consent, the patients will be randomized into two groups: Intervention Group that will perform the PPTHA associated with FES in the gluteus medium; and a Control Group that will perform only the PPTHA.

All patients are evaluated by physiotherapists of Hip Surgery Group of HCPA (HSGHCPA), who helped in the process of randomization, while revaluations are performed at hospital discharge through blinding simple by a researcher linked to the work that will take place only the revaluations and do not have access to the methodological aspects and randomization of the study, the patients are also instructed to not inform what kind of intervention received. The perform assessments are carried out through Amnesia idealized by authors, composed by identification data, history of pathology and current history of previous pathologist. In addition, all patients also underwent the following evaluations: before the intervention and after completion of the interventions, pre hospital discharge.

The evaluation of joint ranges of motion will be carried out through the goniometry which will be performed in accordance with the methodology proposed by Manual Goniometry. Will be assessed by means of goniometry the movements of flexion, extension, adduction, abduction, internal and external rotation of both sides of the hip.

The maximum muscle strength of the gluteus medium will be evaluated through a dynamometer load coupled to a support, stuck to the knee of the patient that will be in lateral decubitus, and will cause the movement of hip extension with both legs. The force shall be measured three times with intervals of 2 minutes of rest between the assessments. The maximum value obtained will be used as voluntary force maximum of the gluteus medium.

Clinical evaluations and functional will be measured by means of the scores of Merle D'aubigne and Postel that has as objective to evaluate the motor performance regarding pain, gait and mobility. The clinical evaluation, the maximum score for pain (total absence), mobility (equal to normal hip) and gear (normal) is 6 and the sum total of the three evaluated areas is 18. The functional assessment the maximum score for pain (no pain) and ability to ambulate (normal) is 12.

The structural adaptations of the gluteus medium from the rehabilitation will be assessed by means of images of ultrasound. For evaluation of muscle architecture will be used a System of portable ultrasound (VIVID i®, GE) with a probe of linear arrangement (60 mm, 7.5 MegaHertz (MHz) - VIVID i®, GE). The portable system will allow the easy scroll for assessment of patients in Inpatient Units. A single researcher is responsible for collection of all images, which are obtained with the muscles at rest. Maps are made in layers of acetate to ensure that images are collected in the same points during the assessments pre and post-training. These images are used in the evaluation of the following parameters of muscle architecture: (1) muscle thickness, which is measured by means of a perpendicular line between the superficial aponeurosis and the deep aponeurosis muscle; (2) length of volume, which represents the length of the muscle fiber and is a parameter that denotes the number of sarcomeres aligned in series and (3) angle of affliction of fibers, obtained by means of the angle formed between the deep aponeurosis and the volume, which is an indication of the size of the muscle fibers (i.e. the number sarcomeres aligned in parallel).

The Control Group receives daily visits of HSGHCPA workouts from PPTHA, already established at HCPA. Already the Intervention Group performs the PPTHA associated with FES during the hospital phase.

ELIGIBILITY:
Inclusion Criteria:

* patients with Coxarthroses Primary and Secondary with THA indication

Exclusion Criteria:

* patients who refused to participate in this study,
* patients with indication for THA by fractures and bone tumors,
* THA review,
* anatomic abnormalities congenital and acquired,
* patients with neurologist lesions that do not understand the commands or with changes in sensitivity in lower limbs
* patients with postoperative infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Anamnesis | The assessment is held a day before the surgery and in the fourth or fifth day in hospital discharge. The time between assessment and reassessment is up to five days.
  Composed of the identification data, history of current and history of Pathology progression of pathologies.

SECONDARY OUTCOMES:
Goniometry | The assessment is held a day before the surgery and in the fourth or fifth day in hospital discharge. The time between assessment and reassessment is up to five days
  Will be performed in accordance with the methodology proposed by Goniometry Manual. Will be assessed by goniometry passive movements of flexion, adduction, abduction, internal and external rotation of the hand operated before and after THA.
Evaluation of muscle strength of gluteus medius | The assessment is held a day before the surgery and in the fourth or fifth day in hospital discharge. The time between assessment and reassessment is up to five days
  Maximum muscle strength of gluteus medius muscle will be evaluated through a portable digital load dynamometer 20 Kilogram force (Kgf), Instrutemp brand, itfg5020 model. With the patient lying supine, the dynamometer is positioned on the underside of the thigh region of the operated limb, next to the patient's knee to score the maximum isometric contraction of abduction and external rotation of the hip, creating a compressive force on the dynamometer. The strength will be measured three times with intervals of 2 minutes of rest between the assessments. The maximum value obtained will be used as the maximum gluteus medius volunteer force.
Functional evaluation of the hip | The assessment is held a day before the surgery and in the fourth or fifth day in hospital discharge. The time between assessment and reassessment is up to five days
  The Harris Hip Score is specific assessment tool designed to assess the results of the ANALYSES, being widely used as a method of comparing the results. Features scale with a maximum of 100 points, including assessment of pain, function,deformity and mobility. Pain and function has the highest weight (44 and 47 points).Range of motion and deformity are of primary importance getting 5 and 4 points respectively. The functionality is subdivided into activities of daily living (14 points) and March (33 points). Total score less than 70 points is considered bad result, 70 to 80 80 to 90 reasonably good and the excellent 100 90.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Umpierres, Master, Principal Investigator — Federal University Rio Grande do Sul
Locations (1):
- Federal University Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No